CLINICAL TRIAL: NCT01525407
Title: Donor Statin Treatment for Prevention of Severe Acute GVHD After Myeloablative Hematopoietic Cell Transplantation
Brief Title: Donor Atorvastatin Treatment for Preventing Severe Acute Graft-Versus-Host Disease in Patients Undergoing Myeloablative Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marco Mielcarek, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2545.00; NCI-2011-03827 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2545.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); R01HL108307 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Atorvastatin; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (donor statin treatment) (Experimental): Donors receive atorvastatin calcium PO beginning on day -14 and continuing until the last day of stem cell collection.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Atorvastatin Calcium; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo myeloablative allogeneic PBSC transplant
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Atorvastatin Calcium — Given PO
  Other Names: CI-981; Lipitor
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo myeloablative allogeneic PBSC transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation

SUMMARY:
This phase II trial studies donor atorvastatin treatment for the prevention of severe acute graft-versus-host disease (GVHD) in patients undergoing myeloablative peripheral blood stem cell (PBSC) transplantation. Giving chemotherapy and total-body irradiation (TBI) before a donor PBSC transplant helps stop the growth of cancer cells. It may also prevent the patient's immune system reject the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving atorvastatin to the donor before transplant may prevent this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether 2 weeks of donor statin treatment reduces the risk of severe acute GVHD.

SECONDARY OBJECTIVES:

I. To assess whether 2 weeks of statin treatment of normal PBSC donors is feasible, tolerable and safe.

OUTLINE:

Donors receive atorvastatin orally (PO) beginning on day -14 and continuing until the last day of stem cell collection.

ELIGIBILITY:
Inclusion Criteria:

* Human leukocyte antigen (HLA)-identical sibling donor
* Myeloablative preparative regimen (i.e., >= TBI 12.0 Gy, >= busulfan (BU) 8.0 mg/kg PO, >= BU 6.4 mg/kg intravenously (IV), >= treosulfan 42 g/m^2 IV) according to investigational study or standard treatment plan; other "myeloablative" preparative regimens are acceptable as long as they are approved by the principal investigator or designee
* Transplantation of PBSC
* Cyclosporine (CSP)-based postgrafting immunosuppression
* Willingness to give informed consent
* DONOR: Age >= 18 years
* DONOR: HLA genotypically identical sibling
* DONOR: Willingness to give informed consent

Exclusion Criteria:

* Nonmyeloablative preparative regimen
* Participation in an investigational study that has acute GVHD as the primary endpoint
* The allogeneic PBSC donor has a contraindication to statin treatment
* DONOR: Age < 18 years
* DONOR: Active liver disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] levels > 2 times the upper limit of normal [ULN])
* DONOR: History of myopathy
* DONOR: Hypersensitivity to atorvastatin
* DONOR: Pregnancy
* DONOR: Nursing mother
* DONOR: Current serious systemic illness
* DONOR: Concurrent treatment with strong inhibitors of hepatic cytochrome P450 (CYP) 3A4 (i.e. clarithromycin, erythromycin, protease inhibitors, azole antifungals)
* DONOR: Current use of statin drug
* DONOR: Failure to meet Fred Hutchinson Cancer Research Center (FHCRC) or local criteria for stem cell donation
* DONOR: Total creatinine kinase > 2 times the ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Stanford University Hospitals and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Donors: Donors receive atorvastatin calcium PO beginning on day -14 and continuing until the last day of stem cell collection.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo myeloablative allogeneic PBSC transplant
  Atorvastatin Calcium: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo myeloablative allogeneic PBSC transplant
- Patients: Recipients of donor stem cells.
Period: Overall Study
Arm/Group | Donors | Patients
Started | 41 | 42
Completed | 38 | 38
Not Completed | 3 | 4
Not completed — Change in recipient treatment plan | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Transplant was delayed | 0 | 1
Not completed — Delay in Transplant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donors | Patients | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Median (Full Range); unit: years] | 54 [22 to 64] | 52 [24 to 69] | 53 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 27 | 55
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Grade 3-4 Acute GVHD
Description: Cumulative incidence rate of grade 3-4 acute GVHD with death as a completing risk, assessed at day 100 in the patients/recipients.
Time Frame: First 100 days after transplant
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.21 [0.10 to 0.35]

2. Secondary Outcome: Chronic Extensive GVHD
Description: Cumulative incidence rate of chronic extensive GVHD with death as a competing risk, assessed at 2 years in the patients/recipients.
Time Frame: 2 years post transplant
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.51 [0.33 to 0.66]

3. Secondary Outcome: Disease-free Survival
Description: Evaluated as Kaplan-Meier estimate in the patients/recipients.
Time Frame: 1 year after transplant
Measure: Number (95% Confidence Interval); unit: disease free survival probability
Arm/Group | Patients
Number analyzed (Participants) | 38
disease free survival probability | 0.47 [0.34 to 0.66]

4. Secondary Outcome: Grades II-IV Acute GVHD
Description: Cumulative incidence rate of grades II-IV acute GVHD with death as a competing risk, assessed at 100 days in the patients/recipients.
Time Frame: First 100 days after transplant
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.78 [0.61 to 0.89]

5. Secondary Outcome: Non-relapse Mortality
Description: Cumulative incidence rate of non-relapse mortalities, assessed at day 100 in the patients/recipients.
Time Frame: At day 100
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.13 [0.05 to 0.26]

6. Secondary Outcome: Non-relapse Mortality
Description: Cumulative incidence rate of non-relapse mortalities, assessed at one year in the patients/recipients.
Time Frame: At 1 year after HCT
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.29 [0.15 to 0.44]

7. Secondary Outcome: Overall Survival
Description: Determined and presented as Kaplan-Meier estimates, assessed at 1 year in the patients/recipients.
Time Frame: 1 year after transplant
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Patients
Number analyzed (Participants) | 38
survival probability | 0.55 [0.42 to 0.74]

8. Secondary Outcome: Proportion of Donors Who Have to Discontinue Atorvastatin Because of Toxicity
Time Frame: Until completion of stem cell collection (on average 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Donors
Number analyzed (Participants) | 41
Participants | 3

9. Secondary Outcome: Proportion of Patients Requiring Secondary Systemic Immunosuppressive Therapy
Time Frame: First 100 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 38
Participants | 5

10. Secondary Outcome: Recurrent or Progressive Malignancy
Description: Cumulative incidence rate of recurrent or progressive malignancy with death as a competing risk, assessed at 3 years in the patients/recipients.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Patients
Number analyzed (Participants) | 38
probability | 0.27 [0.14 to 0.42]

ADVERSE EVENTS:
Time Frame: Donor: SAEs, AEs (≥ grade 2) and UPs will be monitored and recorded from the time the donor starts atorvastatin therapy through the time of discharge from the transplant center after donation of stem cells or 7 days after the discontinuation of the medication, whichever occurs earlier. Recipient: SAEs and UPs (life-threatening or fatal) will be monitored and recorded from the time the recipient starts conditioning therapy through day 100 or discharge from the center, whichever occurs earlier.
Groups:
- Patient Adverse Events: Recipient: SAEs and UPs (life-threatening or fatal) will be monitored and recorded from the time the recipient starts conditioning therapy through day 100 or discharge from the center, whichever occurs earlier.
- Donor Adverse Events: Donor: SAEs, AEs (≥ grade 2) and UPs will be monitored and recorded from the time the donor starts atorvastatin therapy through the time of discharge from the transplant center after donation of stem cells or 7 days after the discontinuation of the medication, whichever occurs earlier.
Arm/Group | Patient Adverse Events | Donor Adverse Events
Serious Adverse Events (participants affected / at risk) | 21/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Adverse Events (N=38) | Donor Adverse Events (N=41)
DAH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 2 (2) | 0 (0)
Fever/Infection (Infections and infestations) | 9 (11) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumotosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GVHD (Immune system disorders) | 7 (8) | 0 (0)
Relapse (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dehydration (Vascular disorders) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
EBV-PTLD (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes